CLINICAL TRIAL: NCT00856180
Title: Pilot Study of Sequential Angiogenic Blockade for the Treatment of Recurrent Mullerian Malignancies
Brief Title: Sequential Angiogenic Blockade for the Treatment of Recurrent Mullerian Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Ursula A. Matulonis, MD, Medical Oncologist, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-148
Record Dates: First submitted 2009-02-25; First posted 2009-03-05 (Estimated); Results first posted 2016-05-17 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: avastin; bevacizumab; cyclophosphamide; cytoxan; mullerian malignancies
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Bevacizumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab then Cyclophosphamide with Bevacizumab (Experimental): Patients were given a regimen of sequential antiangiogenic blockade and disease assessed serologically and radiologically every 2 cycles/6 weeks. Patients started with bevacizumab 15 mg/kg IV every 3 weeks until they experienced progressive disease (PD) [RECIST 1.0 or Rustin criteria] or significant toxicity. If clinically stable as assessed by their treating physician, patients then received cyclophosphamide 50 mg orally (PO) daily continuously with bevacizumab treatment. If second PD occurred, patients discontinued the combination treatment.
  Interventions: Drug: Bevacizumab; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin
Drug: Cyclophosphamide
  Other Names: cytoxan

SUMMARY:
The goals of this study were to evaluate the efficacy and safety of sequentially blocking the angiogenesis pathway via known antiangiogenic mechanisms, first with bevacizumab and then addition of oral cyclophosphamide upon progression of cancer through bevacizumab. The drugs used in this study were chosen because of their known antiangiogenic properties, tolerability, and anti-ovarian cancer effects.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the efficacy of a sequential antiangiogenic blockade regimen of bevacizumab then cyclophosphamide with bevacizumab at disease progression in patients with recurrent ovarian cancer as measured by the proportion of patients who remain on study at three months (4 cycles)
* Assess the safety profile with respect to gastrointestinal perforations

Secondary

* Assess other toxicity/ safety profile of this metronomic antiangiogenic approach
* Assess preliminary response rate and proportion of patients on study at 6 months
* Assess progression-free survival, time to progression and overall survival

Correlative

* Determine if biological correlates of angiogenesis are altered by the addition of sequential therapy
* Determine if changes in biological markers are correlated with clinical state of cancer
* Determine whether biomarkers of angiogenesis can predict and measure response
* Determine whether oncogenic mutations predict response
* Determine whether hypertension and urinary biomarkers such as varying levels of albuminuria predict response to bevacizumab
* Determine patient risk factors for hypertension and proteinuria as toxicities of bevacizumab

STATISTICAL DESIGN:

This study used a two-stage design to evaluate safety and efficacy of sequential antiangiogenic blockade with a regimen of bevacizumab then cyclophosphamide added at disease progression. Safety was measured by the incidence of grade 3-5 gastrointestinal perforation (GIP) during the first 3 months of therapy and efficacy by completion of at least 3 months of therapy. The sample size was determined based on efficacy with the null and alternative therapy completion rate of 50% and 80%, respectively. If 6 or more patients enrolled in the stage one cohort (n=9 patients) completed at least 3 months of therapy then accrual would proceed to stage two (n=11 patients) if there were fewer than 2 cases of grade 3-5 GIP. There was 0.75 probability of stopping the trial at stage one if the true therapy completion rate was 50%. If 13 or fewer patients remained on therapy for at least 3 months by the end of stage two, this regimen would be deemed ineffective. The power to reject the null hypothesis with a one-sided binomial test was 87% assuming 5% significance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.
* Recurrent cancer and have received and failed a previous platinum-based chemotherapy regimen.
* Up to 2 prior lines of chemotherapy in the recurrent setting (either platinum-based or non-platinum regimens). Biologic therapies count as a prior line but hormonal therapies do not count.
* Platinum-resistant or platinum-sensitive recurrence.
* Must be able to take oral medications and have no evidence of bowel obstruction or partial bowel obstruction
* Measurable disease by either RECIST or Rustin criteria
* No chemotherapy, radiation therapy, nor biologic therapy within the last three weeks prior to initiating therapy
* ECOG score of 0 or 1
* Life expectancy of 12 weeks or greater
* 18 years of age or older
* Laboratory values as outlined in the protocol
* Patients with treated limited stage basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the breast or cervix are eligible. Subjects with stage I or II cancer treated with curative intent and no evidence of recurrent disease are also eligible.
* No evidence of preexisting hypertension. If patient has hypertension, it must be controlled medically (less than 150/90) prior to starting bevacizumab
* Normal blood coagulation parameters
* No prior treatment with any other antiangiogenic agents or cyclophosphamide
* For patients who have received prior doxorubicin or pegylated doxorubicin, LVEF must be 50% or greater.

Exclusion Criteria:

* Current, recent (within 4 weeks of the first study infusion), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Active malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within last five years
* Uncontrolled diarrhea
* Prior history of hypertensive crisis or hypertensive encephalopathy
* NYHA Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to day 1
* Known CNS disease, except for treated brain metastasis
* Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS: Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to day 1 will be excluded.
* Significant vascular disease within 6 months prior to day 1
* History of hemoptysis within 1 month prior to day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a UPC ratio of 1.0 or greater at screening
* Known hypersensitivity to any component of bevacizumab
* Pregnancy (positive pregnancy test) or lactation. Use of effective means of contraception (men and women) in subjects of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Matulonis, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Matulonis UA, Pereira L, Liu J, Lee H, Lee J, Whalen C, Campos S, Atkinson T, Hill M, Berlin S. Sequential bevacizumab and oral cyclophosphamide for recurrent ovarian cancer. Gynecol Oncol. 2012 Jul;126(1):41-6. doi: 10.1016/j.ygyno.2012.04.003. Epub 2012 Apr 6. PMID 22487536

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 patients were enrolled between March 2009 and October 2009.
Groups:
- Bevacizumab Then Cyclophosphamide With Bevacizumab: Patients were given a regimen of sequential antiangiogenic blockade and disease assessed serologically and radiologically every 6 weeks. Patients started with bevacizumab 15 mg/kg IV every 3 weeks until they experienced progressive disease (PD) [RECIST 1.0 or Rustin criteria] or significant toxicity. If clinically stable as assessed by their treating physician, patients then received cyclophosphamide 50 mg orally (PO) daily continuously with bevacizumab treatment. If second PD occurred, patients discontinued the combination treatment.
Period: Overall Study
Arm/Group | Bevacizumab Then Cyclophosphamide With Bevacizumab
Started | 20
Completed | 0
Not Completed | 20
Not completed — Adverse Event | 4
Not completed — Progressive Disease | 16

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab Then Cyclophosphamide With Bevacizumab
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 64 [44 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Therapy Completion Rate
Description: The therapy completion rate is defined as the proportion of participants who completed at least 3 months/4 cycles of therapy. Participants were treated until disease progression on the combination regimen or unacceptable toxicity. Clinical response was evaluated based on RECIST 1.0 criteria for measurable disease (MD) participants and Gynecologic Cancer Intergroup (GCIG) CA-125 (Rustin) criteria for non-MD participants. Per RECIST 1.0 for target lesions, PD is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or appearance of new lesions. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Serologic PD is rise in CA-125 or previously normal CA125 that rises to >/=2xULN documented, both requiring 2nd confirmation.
Time Frame: Serologic and radiologic disease assessments occurred every 2 cycles/6 weeks on treatment. Median treatment duration for this study cohort was 7.5 months (range 0.7-20.7).
Population: The analysis dataset is comprised of all treated participants.
Measure: Number (80% Confidence Interval); unit: proportion of participants
Arm/Group | Bevacizumab Then Cyclophosphamide With Bevacizumab
Number analyzed (Participants) | 20
proportion of participants | .75 [0.59 to 0.88]

2. Primary Outcome: Grade 3-5 Gastrointestinal Perforation
Description: All grade 3-5 gastrointestinal perforation events based on CTCAEv3 as reported on case report forms.
Time Frame: Assessed each cycle/3 weeks throughout treatment from time of first dose and up to day 30 post-treatment. Median treatment duration for this study cohort was 7.5 months (range 0.7-20.7).
Population: The analysis dataset is comprised of all treated participants.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Bevacizumab Then Cyclophosphamide With Bevacizumab
Number analyzed (Participants) | 20
proportion of participants | 0.05 [0.003 to .22]

3. Secondary Outcome: Clinical Benefit Response Rate
Description: Clinical benefit response rate is defined as the proportion of participants who achieve confirmed stable disease (SD) or better on treatment based on RECIST 1.0 criteria. Per RECIST 1.0 for target lesions, complete response (CR) is disappearance of all target lesions and partial response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Progressive disease (PD) is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started. SD is neither PR nor PD. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Radiologic disease assessments occurred every 2 cycles/6 weeks on treatment. Median treatment duration for this study cohort was 7.5 months (range 0.7-20.7).
Population: The analysis dataset is comprised of all treated participants.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Groups:
- Platinum Sensitive: At baseline, participants were classified as platinum sensitive or platinum resistant. Platinum sensitive is defined as having had a >6 month interval since last receiving platinum therapy prior to disease recurrence.
- Platinum Resistant: At baseline, participants were classified as platinum sensitive or platinum resistant. Platinum resisistant is defined as having had a </=6 month interval since last receiving platinum therapy prior to disease recurrence.
Arm/Group | Platinum Sensitive | Platinum Resistant
Number analyzed (Participants) | 6 | 14
proportion of participants | 1.00 [0.61 to 1.00] | 0.64 [0.39 to 0.85]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS estimated using Kaplan-Meier methods is defined as the duration of time from the start of bevacizumab alone to documented disease progression (PD) requiring removal from the study or death. If participant ultimately received both bevacizumab and cyclophosphamide then it was the time until PD on both agents. Per RECIST 1.0 for target lesions, PD is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or appearance of new lesions. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Serologic PD is rise in CA-125 or previously normal CA-125 that rises to >/=2xULN documented, both requiring 2nd confirmation. Participants who were event-free were censored at the date of their last disease evaluation.
Time Frame: Radiologic disease assessments occurred every 2 cycles/6 weeks on treatment and every 3 months in follow-up until PD, death or lost to follow-up. Median treatment duration was 7.5 months (range 0.7-20.7) and survival follow-up 23 months..
Population: The analysis dataset is comprised of all treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Then Cyclophosphamide With Bevacizumab
Number analyzed (Participants) | 20
months | 8.41 [2.83 to 15.41]

5. Secondary Outcome: Overall Survival (OS)
Description: OS estimated using Kaplan-Meier methods is defined as the time from study entry to death or date last known alive.
Time Frame: Participants were followed long-term for survival every 3 months from the end of treatment until death or lost to follow-up. Median follow-up was 23 months in this study cohort.
Population: The analysis dataset is comprised of all treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Then Cyclophosphamide With Bevacizumab
Number analyzed (Participants) | 20
months | 22.72 [15.44 to 30.95]

ADVERSE EVENTS:
Time Frame: Assessed each cycle/ 3 weeks throughout treatment from time of first dose and up to day 30 post-treatment.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | Bevacizumab Then Cyclophosphamide With Bevacizumab
Serious Adverse Events (participants affected / at risk) | 14/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab Then Cyclophosphamide With Bevacizumab (N=20)
Cardiac-ischemia (Cardiac disorders) | 1
Obstruction, colon (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Head/headache (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab Then Cyclophosphamide With Bevacizumab (N=20)
Infection Gr0-2 neut, upper airway (Infections and infestations) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Cardiac-other (Cardiac disorders) | 1
Dry eye syndrome (Eye disorders) | 1
Eye, pain (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5
Enteritis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Abdomen, pain (Gastrointestinal disorders) | 2
Stomach, pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 16
Edema head and neck (General disorders) | 1
Edema limb (General disorders) | 2
Leukocytes (Investigations) | 3
Neutrophils (Investigations) | 3
Platelets (Investigations) | 2
ALT, SGPT (Investigations) | 1
AST, SGOT (Investigations) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Joint-function (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 3
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 2
Joint, pain (Musculoskeletal and connective tissue disorders) | 8
Muscle, pain (Musculoskeletal and connective tissue disorders) | 3
Neck, pain (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 2
Head/headache (Nervous system disorders) | 6
Urinary hemorrhage NOS (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 4
Vagina, hemorrhage (Reproductive system and breast disorders) | 1
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 3
Skin-other (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No